CLINICAL TRIAL: NCT06547892
Title: Use of Vasopressin in Patients at High Risk of Acute Kidney Injury Admitted to the ICU: a Feasibility Randomized Clinical Trial
Brief Title: Use of Vasopressin in Patients at High Risk of Acute Kidney Injury Admitted to the ICU
Acronym: NOVA-AKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOVA-AKI
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: Clinical, multicenter, placebo-controlled, double-blind, randomized and feasibility trial with a proposal to include 60 patients in 3 to 4 research centers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization list will be generated with appropriate software, in blocks of 4, by a statistician not involved in patient care. There will be stratification by center. Randomization confidentiality will be guaranteed by central randomization via REDCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vasopressin (Experimental): To dilute vasopressin, an ampoule containing 20 IU/ml (1 ml) of vasopressin will be used, which will be mixed with 100 ml of 0.9% physiological solution, resulting in a solution with a concentration of 0.2 IU/ ml. In this study, both central and peripheral vein infusion will be permitted.
  The vasopressin administration protocol will consist of an initial dose of 0.02 IU/min (equivalent to 6 ml/h), which can be increased to 0.03 IU/min (9 ml/h) if the mean arterial pressure (MAP) is less than or equal to 65 mmHg. On the other hand, if MAP exceeds 90 mmHg, the dose can be reduced to 0.01 IU/min (3 ml/h). The minimum period for adjusting the drug dosage should be one hour.
  In the event that a MAP exceeds 100 mmHg persists, the dose of the drug can be reduced more quickly or even stopped. The duration of vasopressin therapy will be maintained for 7 days, discharge from the ICU, initiation of renal replacement therapy or until death, whichever occurs first.
  Interventions: Drug: Vasopressin
- Placebo (Placebo Comparator): Similar to the intervention protocol, but using a placebo composed of 0.9% saline solution.
  Interventions: Other: 0,9% saline solution

INTERVENTIONS:
Drug: Vasopressin — To dilute vasopressin, an ampoule containing 20 IU/ml (1 ml) of vasopressin will be used, which will be mixed with 100 ml of 0.9% physiological solution, resulting in a solution with a concentration of 0.2 IU/ ml. In this study, both central and peripheral vein infusion will be permitted.
  The vasopressin administration protocol will consist of an initial dose of 0.02 IU/min (equivalent to 6 ml/h), which can be increased to 0.03 IU/min (9 ml/h) if the mean arterial pressure (MAP) is less than or equal to 65 mmHg. On the other hand, if MAP exceeds 90 mmHg, the dose can be reduced to 0.01 IU/min (3 ml/h). The minimum period for adjusting the drug dosage should be one hour.
  Arms: Vasopressin
Other: 0,9% saline solution — Similar to the intervention protocol, but using a placebo composed of 0.9% saline solution.
  Arms: Placebo

SUMMARY:
Renal dysfunction is a frequent complication in patients admitted to intensive care units (ICUs), associated with high morbidity and mortality. Current therapeutic options to prevent this condition are limited and lack robust scientific evidence. This pilot study consists of a multicenter, blinded, randomized clinical trial, unprecedented in the literature to date, aiming to fill this knowledge gap and offer new therapeutic perspectives to improve renal outcomes in critically ill patients admitted to the ICU.

DETAILED DESCRIPTION:
This is a multicenter, placebo-controlled, double-blind, randomized feasibility clinical trial with a proposal to include 60 patients across 3 to 4 research centers.

This study will be conducted in Brazilian hospitals, covering both public and private healthcare profiles across various states of Brazil. Most of these hospitals are academic and teaching institutions, ensuring a wide diversity of data and perspectives for the research.

The objective of this study is to assess the feasibility of conducting a larger subsequent trial to analyze whether the use of vasopressin in patients prone to developing acute kidney dysfunction after admission to intensive care units (ICUs) can prevent the condition (acute kidney dysfunction).

This study is based on the null hypothesis (H0) that there will be no significant difference in the development of acute kidney injury between the group treated with vasopressin and the control group, while the alternative hypothesis (H1) proposes that the administration of vasopressin may reduce the risk of acute kidney injury in high-risk patients admitted to ICUs. The primary objective is to evaluate the feasibility of the study, specifically adherence to the established protocol and the monitoring of potential adverse effects during its conduct.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old);
* Admitted to intensive care units;
* Predicted risk of acute kidney injury calculated based on clinical and laboratory data at ICU admission and is considered eligible if the value in the calculator is equal or greater than 5 points;

Exclusion Criteria:

* Time since admission to the ICU greater than 24 hours;
* Use of vasopressors at the time of inclusion;
* MAP >90 mmHg;
* Hyponatremia (<130 mmol/L);
* Severe TBI with Glasgow Coma Scale < 8;
* Elective surgeries;
* Dialysis chronic kidney disease or acute kidney injury who received renal replacement therapy upon admission or are expected to receive renal replacement therapy within the next 24 hours;
* Suspected or confirmed acute mesenteric ischemia;
* Prospect of death in less than 24 hours;
* Medical team not committed to full investment at the time of inclusion;
* Prior inclusion in the study;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Defined by the inclusion of 60 patients in 3 or more ICUs over a period of 6 months

SECONDARY OUTCOMES:
Creatinine, in mg/dL | 7 days
  Creatinine will be defined by laboratory analysis

OTHER OUTCOMES:
Mortality | 30 days
  Mortality will be defined by medical records

CONTACTS AND LOCATIONS:
Overall Officials: Matheus Silva, Principal Investigator — Hospital do Coracao
Locations (1):
- Matheus Liguori Feliciano da Silva, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Our data dissemination plan will follow the rules of the research institute (Hcor)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 20 months